CLINICAL TRIAL: NCT01571947
Title: Acute Effects of Dietary Fats and Carbohydrate on Insulinaemia, Lipaemia, Inflammatory Responses and Gastrointestinal Peptide Secretion in Subjects With Metabolic Syndrome
Brief Title: Acute Effects of Dietary Fats and Carbohydrate in Subjects With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: A003.11
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Metabolic Syndrome
Keywords: Insulinaemia; inflammatory markers; gastrointestinal peptides; SFA; dietary fats; carbohydrate; insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SFA (Active Comparator)
  Interventions: Other: Acute Effects of Fats and Carbohydrate
- MUFA (Active Comparator)
  Interventions: Other: Acute Effects of Fats and Carbohydrate
- PUFA (Active Comparator)
  Interventions: Other: Acute Effects of Fats and Carbohydrate
- CARB (Active Comparator)
  Interventions: Other: Acute Effects of Fats and Carbohydrate

INTERVENTIONS:
Other: Acute Effects of Fats and Carbohydrate — Test meals were served in the form of muffin + milkshake. For high fat meals, 55g of test fat will be incorporated in muffins, whereas 22g of fat for low fat or high carbohydrate test meal. During study day, subjects were to consume the allocated test meal within 10 minutes.

SUMMARY:
There is increasing evidence suggests that elevated levels of postprandial triacylglycerol (TAG)-rich lipoproteins may promote the development of cardiovascular diseases (CVD). A prolonged and elevated postprandial lipemia is associated with increased risk of CVD by a variety of mechanisms such as insulin resistance, inflammation, endothelial dysfunction and oxidative stress. However, current evidence on the acute effects of type of fats on postprandial insulinaemia, gastrointestinal peptide secretion, inflammatory response, as well as satiation are limited and inconsistent, in particular in metabolic syndrome population in Asian. Hence, this study aimed to investigate the postprandial effects of high fat meals enriched with i) palm olein, ii) high oleic sunflower oil, and iii) high linoleic sunflower oil, compared with a low fat/high carbohydrate meal, in 30 subjects with metabolic syndrome.

DETAILED DESCRIPTION:
A randomized, double-blind, crossover design study was conducted to test the acute effects of high fat meals enriched with (1) saturated fatty acids (SFA); (2) monounsaturated fatty acids (MUFA); (3) polyunsaturated fatty acids (PUFA) vs. (4) a low fat/high carbohydrate (CARB) meal on postprandial insulinaemic, lipaemic and inflammatory responses, as well as gastrointestinal peptide secretion and satiation on 30 metabolic syndrome subjects (15 men and 15 women). Primary outcome of this study is postprandial changes of C-peptide. Other measured outcomes including insulin and glucose responses, lipids, cytokines and gastrointestinal peptides. Subjective appetite measurements were taken as exploratory outcomes using visual analogue scales.

Subjects were asked to participate in four postprandial challenges, separated by at least one week. On the day preceding the postprandial intervention, subjects were provided a low fat meal (< 10 g) to consume as their evening meal. They were required to fast over night after 10 pm and arrive at the research unit at 7:30 am - 9:00 am the following morning. Fasting blood samples were collected and subjects were instructed to consume the allocated test meal within 10 minutes. Further venous blood will be collected at regular intervals for up to 6 hours postprandially. During the 6 hours of the experimental study, the subjects were refrained from the consumption of any food or drink except plain water which they will be asked to consume at regular intervals (up to 750 mL over the 6 hours).

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 60
* Elevated TAG with at least 1.7 mmol/L
* Low HDL cholesterol (< 1.04 mmol/L for men, 1.3 mmol/L for women)
* Elevated blood pressure (systolic at least 130, diastolic at least 85 mmHg)
* Increased waist circumference (at least 90cm for men, 80cm for women)
* Fasting plasma glucose between 5.6 and 7.0 mmol/L

Exclusion Criteria:

* Underweight
* Current use of antihypertensive or lipid lowering medication
* Alcohol intake exceeding a moderate intake (> 28 units per week)
* Medical history of myocardial infarction, angina, thrombosis, stroke, cancer or diabetes
* Pregnancy or breast-feeding
* Smoker

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
C-peptide | 6 hours (0, 15, 30, 60, 90, 120, 180, 240, 300 and 360 min)

SECONDARY OUTCOMES:
Insulin | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kim-Tiu Teng, PhD, Principal Investigator — Malaysia Palm Oil Board
Locations (2):
- Malaysia (2):
  - Malaysia Palm oil Board, Kajang, Selangor
  - Malaysian Palm Oil Board (MPOB), Kajang, Selangor

REFERENCES:
- [Derived] Chang CY, Kanthimathi MS, Tan AT, Nesaretnam K, Teng KT. The amount and types of fatty acids acutely affect insulin, glycemic and gastrointestinal peptide responses but not satiety in metabolic syndrome subjects. Eur J Nutr. 2018 Feb;57(1):179-190. doi: 10.1007/s00394-016-1307-9. Epub 2016 Sep 8. PMID 27632019
- [Derived] Teng KT, Chang CY, Kanthimathi MS, Tan AT, Nesaretnam K. Effects of amount and type of dietary fats on postprandial lipemia and thrombogenic markers in individuals with metabolic syndrome. Atherosclerosis. 2015 Sep;242(1):281-7. doi: 10.1016/j.atherosclerosis.2015.07.003. Epub 2015 Jul 7. PMID 26232169